CLINICAL TRIAL: NCT05341349
Title: Safety and Efficacy of SRS and Immune Checkpoint Inhibitors (ICI) Concurrent With NovoTTF-200M in Melanoma Brain Metastases
Brief Title: Stereotactic Radiosurgery and Immune Checkpoint Inhibitors With NovoTTF-200M for the Treatment of Melanoma Brain Metastases
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Cancer Institute (NCI) (NIH); NovoCure Ltd. (Industry)
Responsible Party: Principal Investigator, Mohammad K. Khan, Principal Investigator, Emory University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00003588; NCI-2021-05980 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); RAD5236-21 (Other: Emory University Hospital/Winship Cancer Institute); P30CA138292 (NIH)
Record Dates: First submitted 2022-04-11; First posted 2022-04-22 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Clinical Stage IV Cutaneous Melanoma AJCC v8; Melanoma of Unknown Primary; Metastatic Malignant Neoplasm in the Brain; Metastatic Melanoma; Metastatic Mucosal Melanoma; Metastatic Ocular Melanoma; Pathologic Stage IV Cutaneous Melanoma AJCC v8
MeSH Terms: conditions — Brain Neoplasms; Melanoma; Uveal Melanoma | interventions — Ipilimumab; CTLA-4 Antigen; Nivolumab; pembrolizumab; Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Arm I (SRS, pembrolizumab, TTFields) (Experimental): Patients receive standard of care pembrolizumab and undergo 3-5 fractions SRS. Patients also undergo TTFields over 8 hours daily using NovoTTF-100M device until intra-cranial progression or until end of immunotherapy treatments at the discretion of the treating physician in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Pembrolizumab; Radiation: Stereotactic Radiosurgery; Procedure: Tumor Treating Fields Therapy
- Arm II (nivolumab, ipilimumab, SRS, TTFields) (Experimental): Patients receive standard of care nivolumab and ipilimumab and undergo 3-5 fractions SRS. Patients also undergo TTFields over 8 hours daily using NovoTTF-100M device until intra-cranial progression or until end of immunotherapy treatments at the discretion of the treating physician in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Ipilimumab; Biological: Nivolumab; Radiation: Stereotactic Radiosurgery; Procedure: Tumor Treating Fields Therapy

INTERVENTIONS:
Biological: Ipilimumab — Given IV
  Other Names: Anti-Cytotoxic T-Lymphocyte-Associated Antigen-4 Monoclonal Antibody; BMS-734016; Ipilimumab Biosimilar CS1002; MDX-010; MDX-CTLA4; Yervoy
  Arms: Arm II (nivolumab, ipilimumab, SRS, TTFields)
Biological: Nivolumab — Given IV
  Other Names: BMS-936558; CMAB819; MDX-1106; NIVO; Nivolumab Biosimilar CMAB819; ONO-4538; Opdivo
  Arms: Arm II (nivolumab, ipilimumab, SRS, TTFields)
Biological: Pembrolizumab — Given IV
  Other Names: Keytruda; Lambrolizumab; MK-3475; SCH 900475
  Arms: Arm I (SRS, pembrolizumab, TTFields)
Radiation: Stereotactic Radiosurgery — Undergo SRS
  Other Names: Stereotactic External Beam Irradiation; stereotactic external-beam radiation therapy; Stereotactic Radiation Therapy; Stereotactic Radiotherapy; stereotaxic radiation therapy; stereotaxic radiosurgery
Procedure: Tumor Treating Fields Therapy — Undergo TTFields
  Other Names: Alternating Electric Field Therapy; TTF; TTFields

SUMMARY:
This phase I trial finds out the side effects and possible benefits of stereotactic radiosurgery and immune checkpoint inhibitors with NovoTTF-100M for the treating of melanoma that has spread to the brain (brain metastases). Stereotactic radiosurgery is a type of external radiation therapy that uses special equipment to position the patient and precisely give a single large dose of radiation to a tumor. It is used to treat brain tumors and other brain disorders that cannot be treated by regular surgery. Immunotherapy with monoclonal antibodies, such as pembrolizumab, nivolumab and ipilimumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. NovoTTF-100M is a portable battery operated device which produces tumor treating fields in the body by means of surface electrodes placed on the skin. Tumor treating fields are low intensity, intermediate frequency electric fields that pulse through the skin to disrupt cancer cells' ability to divide. Giving stereotactic radiosurgery and immune checkpoint inhibitors with NovoTTF-100M may work better than stereotactic radiosurgery and immune checkpoint inhibitors.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the safety of combining tumor treating fields therapy (TTFields) to the two therapeutic backbones (stereotactic radiosurgery [SRS]+pembrolizumab and SRS+dual-checkpoint).

SECONDARY OBJECTIVES:

I. To evaluate skin toxicity (grade 1 & 2 skin > 20% and grade 3 & 4 toxicity above 2% at 4-6 weeks and 3 months). (Skin AES include Dermatitis, Erosions, Infections, Ulceration).

II. Control of the treated lesion in the brain with SRS+ immune checkpoint inhibitors (ICI) (i.e. local control), development of additional sites of disease in the brain that were not initially treated with SRS (i.e. anywhere intra-cranial failure), intra-cranial progression free survival (local control of the area that received SRS and anywhere intra-cranial failure), extra-cranial disease response (overall progression free survival), and overall survival.

III. To evaluate treatment response at un-irradiated and extra-cranial sites (i.e. the abscopal effect) with all three arms.

IV. To compare differences in potential serological and immune biomarkers, pretreatment, during treatment, and post treatment.

V. Symptomatic radionecrosis rates at 3 and 6 months.

OUTLINE: Patients are assigned to 1 of 2 arms.

ARM I: Patients receive standard of care pembrolizumab and undergo 3-5 fractions SRS. Patients also undergo TTFields over 8 hours daily using NovoTTF-100M device until intra-cranial progression or until end of immunotherapy treatments at the discretion of the treating physician in the absence of disease progression or unacceptable toxicity.

ARM II: Patients receive standard of care nivolumab and ipilimumab and undergo 3-5 fractions SRS. Patients also undergo TTFields over 8 hours daily using NovoTTF-100M device until intra-cranial progression or until end of immunotherapy treatments at the discretion of the treating physician in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 28 days.

ELIGIBILITY:
Inclusion Criteria:

* Be willing and able to provide written informed consent for the trial
* Have diagnosis of malignant melanoma.
* Be >= 22 years of age on the day of signing informed consent
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0-1 or Karnofsky performance status >= 70%
* Patients must have histological diagnosis of melanoma
* Preference is for treatment naive patients that have not gotten previous immunotherapy. However, if approved by principal investigator (PI), patients that have gotten prior PD1 and/or dual immune checkpoint inhibitor therapy may be allowed on this trial if they have progressed intra-cranially or extra-cranially, and have very limited disease progression.
* Patient must be asymptomatic at time of getting SRS (day 0) on trial. Prednisone =< 20 mg/day (4 mg or less of dexamethasone equivalent) for at least 7 days prior to treatment is allowed
* Patients with ocular, mucosal and unknown primary melanoma will also be eligible
* Patients with 1-10 untreated brain metastases at time of initial brain metastases diagnosis (surgery to at least one of the brain lesions and/or biopsy of a lesion for diagnostic purposes and/or for standard of care purposes is acceptable). If patient has surgical removal of at least one lesion, the investigator would wait for a reasonable time after surgery to start the TTFields, SRS and Immunotherapy. This is typically around 2-4 weeks after resection and clearance by neurosurgery to start the treatment. However, the exact time to start would depend on institutional standard of care practice pattern. Enrollment of patient can take place before or after planned surgery.
* Eligible for hypofractionation approach (9 Gy x 3 or 6 Gy x 5). 9 Gyx 3 is preferred approach, but 6 Gy x 5 fractions is acceptable
* Eligible for immunotherapy and TTFields. The TTField wires will be removed immediately before the SRS delivery and then reconnected again immediately after SRS each session. The arrays will be left on the skin during SRS. This is to minimize any electrical discharge from the wires that may occur as a result of SRS beams going through the arrays and/or lead to any dose heterogeneity during SRS delivery and/or damage the electrical, battery operated equipment
* Be willing to comply with NovoTTF-100M device treatment for at least 75% of the time
* Must have caregiver or self support available to assist transducer array exchange.
* Prior radiation to the primary and/or regional radiotherapy for melanoma is acceptable.
* Baseline labs as within standard of care (complete blood count [CBC], comprehensive metabolic panel [CMP], lactate dehydrogenase [LDH], erythrocyte sedimentation rate [ESR], etc) are required within 28 days of enrollment.
* Have at least one measurable extra-cranial site of disease
* Patients must have at least 14 days to recover from all prior treatment, including surgery, chemotherapy, immunotherapies, prior to enrollment on this protocol.
* Absolute neutrophil count (ANC) >= 1,500 /mcL (performed within 28 days of treatment initiation)
* Platelets >= 100,000 / mcL (performed within 28 days of treatment initiation)
* Hemoglobin >= 9 g/dL or >= 5.6 mmol/L without transfusion or erythropoietin (EPO) dependency (within 7 days of assessment) (performed within 28 days of treatment initiation)
* Serum creatinine =< 1.5 X upper limit of normal (ULN) OR measured or calculated creatinine clearance (glomerular filtration rate [GFR] can also be used in place of creatinine or creatinine clearance [CrCl]) >= 60 mL/min for subject with creatinine levels > 1.5 X institutional ULN (performed within 28 days of treatment initiation)
* Serum total bilirubin =< 1.5 X ULN OR direct bilirubin =< ULN for subjects with total bilirubin levels > 1.5 ULN
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 X ULN OR =< 5 X ULN for subjects with liver metastases (performed within 28 days of treatment initiation)
* Albumin >= 2.5 mg/dL (performed within 28 days of treatment initiation)
* International normalized ratio (INR) or prothrombin time (PT) =< 1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or partial thromboplastin time (PTT) is within therapeutic range of intended use of anticoagulants (performed within 28 days of treatment initiation)
* Activated partial thromboplastin time (aPTT) =< 1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants (performed within 28 days of treatment initiation)
* Female subject of childbearing potential must have a negative urine or serum pregnancy within 2 weeks prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.

  * Female subjects of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study medication. Subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 2 year. This is referring primarily to the use of immunotherapy.
  * Male subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy. This is referring primarily to the use of immunotherapy.
  * Abstinence is acceptable, if this is the usual life style and preferred contraception for the patient

Exclusion Criteria:

* Implanted electrical device (TTField is not implanted device, but worn externally)
* Sensitive to gel used with electrocardiogram (ECG), electrical nerve stimulation, contact with gel used with Novo-TTF system
* Has a diagnosis of immunodeficiency or is receiving systemic steroids (less than or equal to 20 mg prednisone equivalent or less than 4 mg dexamethasone per day at time of start of treatment is ok) therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment
* If they have brain metastases located in the brain stem (including midbrain, pons, or medulla)
* Inability to undergo MRI evaluation for treatment planning and follow-up
* Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment. Has a diagnosis of immunodeficiency or is receiving systemic steroids (less than or equal to 20 mg prednisone equivalent or 4 mg dexamethasone at time of start of treatment is ok) therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment
* Has a known history of active TB (Bacillus tuberculosis)
* Hypersensitivity to pembrolizumab, ipilimumab or any of its recipients
* Hypersensitivity to hydrogel (needed for TTFields)
* Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study day 1 or who has not recovered (i.e., =< grade 1 or at baseline) from adverse events due to a previously administered agent

  * Note: Subjects with =< grade 2 neuropathy are an exception to this criterion and may qualify for the study
  * Note: If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy
* Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer
* Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment
* Has known history of (non-infectious) pneumonitis that required steroids (less than or equal to 20 mg prednisone equivalent at time of start of treatment is ok) or current pneumonitis
* Has an active infection requiring systemic therapy
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment
* Has a known history of human immunodeficiency virus (HIV) (HIV 1/2 antibodies)
* Has known active hepatitis B (e.g., hepatitis B surface antigen [HBsAg] reactive) or hepatitis C (e.g., hepatitis C virus [HCV] ribonucleic acid [RNA] [qualitative] is detected)
* Has received a live vaccine within 30 days of planned start of study therapy

  * Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist) are live attenuated vaccines, and are not allowed
* Implanted pacemaker, defibrillator, deep brain stimulator, or documented clinically significant arrhythmias
* Evidence of increased intracranial pressure meets any of the follow criteria of raised intracranial pressure:

  * Midline shift > 5 mm
  * Clinically significant papilledema
  * Nausea/vomiting related to raised intracranial pressure
  * Reduced level of consciousness related to raised intracranial pressure

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2022-10-13 (Actual); Primary Completion 2026-03-06 (Estimated); Study Completion 2027-03-06 (Estimated)

PRIMARY OUTCOMES:
The percentage of patients developing grade 3 CNS toxicity | At 3 months
  Will be analyzed separately for arms 1 and 2. Radiation Therapy Oncology Group Grade 3 CNS toxicity will be measured using RTOG grade 3 CNS toxicity and reported as percentage of patients developing grad 3 CNS toxicity. Higher score means more patients developing toxicity. Lower score means less patients developing toxicity.

SECONDARY OUTCOMES:
Rates of skin toxicity | At 4-6 weeks and 3 months
  As measured by Common Terminology Criteria for Adverse Events (CTCAE) 5.0, will be reported using frequencies and percentages. Skin toxicity will be analyzed separately for arms 1 and 2.
Rates of alopecia | At 4-6 weeks and 3 months
  As measured by CTCAE 5.0, will be reported using frequencies and percentages. Alopecia will be analyzed separately for arms 1 and 2.
Time to progression | At 6 and 12 months
  Will be defined as the time without evidence of tumor progression from time of stereotactic radiosurgery (SRS). Local control will be estimated using the Kaplan-Meier method. A 95% confidence interval for 6-month and 12-month local control will be estimated using the Greenwood formula. Local control will be analyzed separately for arms 1 and 2.
Intracranial control | At 6 and 12 months
  Will be defined as the time without evidence of tumor progression from time of SRS. Intracranial control will be estimated using the Kaplan-Meier method. A 95% confidence interval for 6-month and 12-month intracranial control will be estimated using the Greenwood formula. Intracranial control will be analyzed separately for arms 1 and 2.
Progression free survival (PFS) | From SRS to disease progression or death, assessed up to 2 years
  PFS will be estimated using the Kaplan-Meier method, and a 95% confidence interval for median PFS will be estimated using the Brookmeyer-Crowley approach. PFS will be analyzed separately for arms 1 and 2.
Overall survival (OS) | From SRS to death, assessed up to 2 years
  OS will be estimated using the Kaplan-Meier method, and a 95% confidence interval for median OS will be estimated using the Brookmeyer-Crowley approach. OS will be analyzed separately for arms 1 and 2.

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad K Khan, MD, PhD, Principal Investigator — Emory University Hospital/Winship Cancer Institute
Locations (1):
- Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia, United States